CLINICAL TRIAL: NCT00966381
Title: Breastfeeding and Exercise for Healthy Infants and Postpartum Moms Too!
Acronym: BEHIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Greensboro (Other)
Collaborators: North Carolina State Agricultural Research Service (Unknown)
Responsible Party: Principal Investigator, Cheryl A Lovelady, PhD RD, Professor, University of North Carolina, Greensboro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 06-0259
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Results first posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2022-07

CONDITIONS: Osteoporosis; Obesity; Weight Loss
Keywords: breastfeeding; bone mineral density; exercise; diet
MeSH Terms: conditions — Osteoporosis; Obesity; Weight Loss; Breast Feeding; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Other): The minimal care group will receive standard public health information on nutrition from the American Heart Association twice during the 16-week intervention. Upon completion of the endpoint measurement (20 weeks postpartum), they will be given all intervention materials.
  Interventions: Other: Exercise and weight loss intervention
- Exercise Group (Experimental): The intervention group will participate in a 16-week exercise and diet intervention from 4 to 20 weeks postpartum. The PI will travel to the participant's homes three times per week during the 16-week intervention to guide mothers with the exercise program, ensure dietary compliance, and provide social support. The 16-week exercise protocol consists of strength training three times per week and walking 10,000 steps per day at least five days per week.
  Interventions: Other: Exercise and weight loss intervention

INTERVENTIONS:
Other: Exercise and weight loss intervention — randomized control trial, stratified by parity
  Other Names: BH2

SUMMARY:
Approximately 8 million American women suffer from osteoporosis, and one out of every two women over the age of 50 will have an osteoporotic-related fracture in their lifetime (42). While epidemiological studies suggest that pregnancy and lactation are not associated with risk of fractures later in life, these studies did not control for site-specific decrements in bone mineral density (BMD). In addition, 55% of American women between the ages of 20 to 39 are overweight (14). Excess weight retention after pregnancy increases a woman's risk for developing a chronic disease later in life (44). There is a paucity of research on exercise and dietary interventions in postpartum lactating women aimed at promotion of bone health and weight loss.

The goal of this study is to promote long-term lifestyle changes through a home based strength training, aerobic, and nutrition intervention targeting overweight lactating women. The objective is to attenuate lactation-induced bone loss and promote weight loss. We hypothesize that the intervention group will lose a greater amount of fat mass while preserving lean mass and bone mineral mass and increase levels of anabolic hormones through diet and exercise compared to the minimal care group. Additionally, the acquisition of such knowledge is unique since no other studies have measured growth hormone and insulin-like growth factor-1 in lactating women with respect to bone and exercise. This intervention will encourage breastfeeding, weight loss and an increase in bone density resulting in healthy infants and mothers.

The proposed research is the first to examine the effects of a resistance exercise and weight loss intervention on attenuation of lactation-induced bone loss in overweight women. To our knowledge, this is the first study to use MyPyramid for Menu Planner for Moms for dietary counseling using the total diet approach. The expected outcomes are the intervention group will lose weight while preserving lean body mass, bone mineral mass and increase cardiovascular fitness and strength compared to the minimal care group. Additionally, the exercise group will improve the overall quality of their diet using internet based technology. An increase in activity and promotion of weight loss through a modest reduction in calories may lead to overall improvement of the mother's bone and health status later in life.

DETAILED DESCRIPTION:
Participants will be randomized, stratified by parity, into either an intervention or minimal care group after all baseline measurements are complete (3 +/- 1 wk postpartum).

The specific aims of this project are to evaluate in overweight lactating women at 3 and 20 weeks postpartum (PP) whether an exercise and weight loss intervention, compared to a minimal care group, will:

1. Improve body composition. The working hypothesis for this aim is the intervention group will lose less lean body mass and bone mineral mass and promote more fat loss compared to the minimal care group at 20 weeks PP.
2. Promote an increase in cardiovascular fitness and strength. The working hypothesis for this aim is the intervention group will increase predicted maximal oxygen consumption and maximal strength compared to the minimal care group at 20 weeks PP.
3. Affect bone-related hormones. The working hypothesis for this aim is the intervention group will increase growth hormone and insulin-like growth factor-1 compared to the minimal care group at 20 weeks PP.
4. Improve total diet or overall pattern of food eaten. The working hypothesis for this aim, based on menu modeling with MyPyramid (16), is the intervention group will improve the quality of their intake by consuming the recommended amounts of food groups established by MyPyramid compared to the minimal care group at 20 weeks PP.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the study, women must be less than 3 weeks postpartum, between the ages of 23 to 40, with a body mass index (BMI) between 25 and 30 kgm-2), exclusively breastfeeding, sedentary for the past 3 months (< 3 weekly sessions of moderate aerobic activity), non-smokers, medically cleared for exercise by their physician, and agree to randomization.

Exclusion Criteria:

* Exclusion criteria for the study are delivery by cesarean section, have medical complications where exercise is contraindicated, or a disease that would affect hormone levels.

Ages: 23 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl A Lovelady, PhD RD, Principal Investigator — UNC Greensboro
Locations (1):
- UNC-Greensboro, Greensboro, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from physicians' offices and childbirth classes. Recruitment was from 2008-2010.
Groups:
- Control: The minimal care group will receive standard public health information on nutrition from the American Heart Association twice during the 16-week intervention. Upon completion of the endpoint measurement (20 wks postpartum), they will be given all intervention materials.
- Exercise Group: The intervention group will participate in a 16-week exercise and diet intervention from 4 to 20 wks postpartum. The PI will travel to the participant's homes three times per week during the 16-week intervention to guide mothers with the exercise program, ensure dietary compliance, and provide social support. The 16-wk exercise protocol consists of strength training three times per week and walking 10,000 steps per day at least five days per week.
Period: Overall Study
Arm/Group | Control | Exercise Group
Started | 15 | 16
Completed | 13 | 14
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Exercise Group | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (3.8) | 31.9 (3.1) | 31.1 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density-Total Body
Description: The results reported are percent change in total body bone mineral density.
Time Frame: Measured at baseline (4 weeks postpartum) and endpoint (16 weeks postpartum)
Measure: Mean (Standard Deviation); unit: percent change in BMD (g/cm2)
Arm/Group | Control | Exercise Group
Number analyzed (Participants) | 13 | 14
percent change in BMD (g/cm2) | -0.3 (2.4) | -1.1 (0.8)
Statistical Analysis 1: Comparison: Control vs Exercise Group; Test type: Superiority; p < 0.05, ANOVA

2. Primary Outcome: Bone Mineral Density-lumbar Spine
Description: Bone mineral density was measured at the lumbar spine. The results reported are the percent change in bone mineral density.
Time Frame: Measured at baseline (4 weeks postpartum) and endpoint (20 weeks postpartum)
Measure: Mean (Standard Deviation); unit: percent change in BMD (g/cm^2)
Arm/Group | Control | Exercise Group
Number analyzed (Participants) | 13 | 14
percent change in BMD (g/cm^2) | -3.7 (3.3) | -3.4 (2.5)
Statistical Analysis 1: Comparison: Control vs Exercise Group; Test type: Superiority; p < 0.05, ANOVA

3. Secondary Outcome: Body Composition
Description: outcome reported as percent change in percent body fat
Time Frame: measured at baseline (4 weeks postpartum) and endpoint (16 weeks postpartum)
Measure: Mean (Standard Deviation); unit: percentage of change in percent fat
Arm/Group | Control | Exercise Group
Number analyzed (Participants) | 13 | 14
percentage of change in percent fat | -6.8 (8.1) | -8.2 (11.1)
Statistical Analysis 1: Comparison: Control vs Exercise Group; Test type: Superiority; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: Data were collected from baseline to endpoint measurements, which was 5 months.
Arm/Group | Control | Exercise Group
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes